CLINICAL TRIAL: NCT06944431
Title: Application of Continuous Passive Motion to Prevent Ankle Contracture and Muscle Loss in the Mechanically Ventilated Patients
Brief Title: Using Continuous Passive Motion to Prevent Ankle Problems in ICU Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SKH-IRB-20240808R
Record Dates: First submitted 2025-04-16; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Joint Contracture; Mechanical Ventilation; ICU-acquired Weakness; Critical Illness; Muscle Atrophy
Keywords: continuous passive motion; ankle joint contracture; ICU-acquired weakness; mechanical ventilation; ultrasound muscle assessment; critical illness; rehabilitation
MeSH Terms: conditions — Critical Illness; Muscular Atrophy | interventions — Motion Therapy, Continuous Passive

STUDY DESIGN:
Intervention Model Description: This is a within-subject controlled study using a single-group assignment model. Each participant received continuous passive motion (CPM) therapy on the left ankle (intervention side), while the right ankle served as the control without CPM. This design allows for internal comparison within the same individual.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CPM Intervention Group (Experimental): All participants received continuous passive motion (CPM) therapy on the left ankle once daily for 7 consecutive days during mechanical ventilation. The right ankle served as the within-subject control with no intervention. This single-arm study used a within-subject control design.
  Interventions: Device: Continuous Passive Motion (CPM)

INTERVENTIONS:
Device: Continuous Passive Motion (CPM) — Continuous passive motion was applied to the left ankle joint for 60 minutes per day using a motorized CPM device. The therapy was initiated within 48 ho

SUMMARY:
The goal of this clinical trial is to learn if continuous passive motion (CPM) helps prevent ankle joint contracture and muscle loss in critically ill, mechanically ventilated ICU patients. It will also evaluate the feasibility and safety of implementing CPM in this population. The main questions it aims to answer are:

Does CPM help preserve ankle dorsiflexion range of motion during immobilization in the ICU?

Can ultrasound measurements detect changes in tibialis anterior muscle condition in response to CPM?

Researchers will compare one ankle receiving CPM to the other ankle without intervention in the same patient to assess differences in joint mobility and muscle morphology.

Participants will:

Receive CPM therapy on one ankle for 30 minutes, twice daily, over a 7-day period or until ICU discharge

Undergo goniometric and ultrasound assessments at baseline and at the end of the intervention

Remain under usual ICU care and monitoring while enrolled in the study

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥ 18 years
* Admitted to the ICU with acute respiratory failure requiring mechanical ventilation
* Expected to remain mechanically ventilated for at least 7 days
* Sedated and unable to participate in active mobilization
* No contraindications for passive ankle movement
* Informed consent obtained from legal representative

Exclusion Criteria:

* Pre-existing neuromuscular disorders affecting lower limb mobility (e.g., stroke with hemiparesis, myasthenia gravis)
* Recent orthopedic surgery or trauma involving the lower limbs
* Presence of lower limb amputation
* Peripheral vascular disease with critical limb ischemia
* Active deep vein thrombosis in either leg
* Significant wounds, pressure ulcers, or skin breakdown at the heel
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-11-20 (Actual); Primary Completion 2025-02-24 (Actual); Study Completion 2025-03-14 (Actual)

PRIMARY OUTCOMES:
Change in Passive Ankle Dorsiflexion Range of Motion (ROM) | Baseline and Day 7
  Difference in passive ankle dorsiflexion angle between baseline and Day 7, measured using a goniometer. The left (intervention) and right (control) ankles will be compared within each subject. Reported in degrees (°).

SECONDARY OUTCOMES:
Tibialis Anterior Muscle Thickness | Baseline and Day 7
  Change in muscle thickness of the tibialis anterior as measured by ultrasound. Measurements will be obtained directly from B-mode ultrasound images using the built-in caliper function of the ultrasound machine. Values will be reported in centimeters (cm).
Tibialis Anterior Muscle Cross-section Area | Baseline and Day 7
  Change in cross-sectional area of the tibialis anterior muscle as measured by ultrasound. Measurements will be obtained directly using the built-in area tracing tool on the ultrasound machine during B-mode imaging. Values will be reported in square centimeters (cm²).
Tibialis Anterior Muscle Pennation Angle | Baseline and Day 7
  Change in pennation angle of the tibialis anterior muscle as measured from B-mode ultrasound images. Angle will be calculated using ImageJ software from the fascicle orientation relative to the deep aponeurosis. Reported in degrees (°).
Tibialis Anterior Muscle Echointensity | Baseline and Day 7
  Change in echointensity of the tibialis anterior muscle as measured from B-mode ultrasound images. Echointensity will be quantified using ImageJ software as the mean and standard deviation of grayscale values within a manually selected region of interest (ROI), ranging from 0 (black) to 255 (white). Reported in grayscale arbitrary units (AU).

CONTACTS AND LOCATIONS:
Locations (1):
- Shin Kong Wu Ho-su Memorial Hospital, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) will not be shared due to the small sample size and the risk of re-identification, especially in a critically ill ICU population. The study was not designed with data sharing infrastructure in place.

REFERENCES:
- [Derived] Lin CC, Lin YJ, Wang HC, Hsu WC. Continuous passive motion for prevention of ankle contracture and muscle loss in mechanically ventilated ICU patients. BMC Res Notes. 2025 Oct 1;18(1):409. doi: 10.1186/s13104-025-07457-z. PMID 41035043